CLINICAL TRIAL: NCT01920269
Title: Intravesical Adjuvant Electromotive Mitomycin-C in Patients With pTa-pT1 and G1-G2 Non-muscle Invasive Bladder Cancer: a Randomized Controlled Trial
Brief Title: Intravesical Adjuvant Electromotive Mitomycin-C
Acronym: EMDA/MMC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Collaborators: University of L'Aquila (Other); University Of Perugia (Other)
Responsible Party: Principal Investigator, Savino M. Di Stasi, Associate Professor of Urology, MD, PhD, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTV-72-1993
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Bladder Cancer TNM Staging Primary Tumor (T) Ta; Bladder Cancer TNM Staging Primary Tumor (T) T1; Bladder Cancer Transitional Cell Grade
Keywords: non-muscle invasive bladder cancer; intravesical chemotherapy; mitomycin; passive diffusion; electromotive drug administration
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Transurethral resection alone (Active Comparator): Patients underwent urinary cytology, random cold-cup biopsies of the bladder and prostatic urethra-ie, and complete transurethral resection of all bladder tumour visible on endoscopy, ensuring muscle is included in resected samples. Response to treatment will be assessed with cystoscopy, biopsy and urinary cytology at 3-month intervals for 2 years, 6-month intervals for 3 years and yearly thereafter.
  Interventions: Procedure: Trans-urethral resection
- Intravesical passive diffusion mitomycin (Active Comparator): Patients underwent urinary cytology, random cold-cup biopsies of the bladder and prostatic urethra, and complete transurethral resection of all bladder tumour visible on endoscopy, ensuring muscle is included in resected samples. Patients are scheduled to receive an initial 6 intravesical mitomycin treatments at weekly intervals commencing 2 weeks after endoscopic procedures. Patients are placed on fluid restriction and oral sodium bicarbonate before intravesical mitomycin treatments. Patients who have a complete response to the initial 6 weekly treatments underwent a further 10 monthly instillations. Response to treatment will be assessed with cystoscopy, biopsy and urinary cytology at 3-month intervals for 2 years, 6-month intervals for 3 years and yearly thereafter.
  Interventions: Procedure: Trans-urethral resection; Drug: intravesical passive diffusion mitomycin
- Intravesical electromotive mitomycin (Active Comparator): Patients underwent urinary cytology, random cold-cup biopsies of the bladder and prostatic urethra, and complete transurethral resection of all bladder tumour visible on endoscopy, ensuring muscle is included in resected samples. Patients are scheduled to receive an initial 6 intravesical mitomycin treatments at weekly intervals commencing 2 weeks after endoscopic procedures. Patients are placed on fluid restriction and oral sodium bicarbonate before intravesical mitomycin. Patients who have a complete response to the initial 6 weekly treatments underwent a further 10 monthly instillations. Response to treatment will be assessed with cystoscopy and urinary cytology at 3-month intervals for 2 years, 6-month intervals for 3 years and yearly thereafter.
  Interventions: Procedure: Trans-urethral resection; Drug: intravesical passive diffusion mitomycin; Device: intravesical electromotive mitomycin

INTERVENTIONS:
Procedure: Trans-urethral resection — Patients underwent urinary cytology of the bladder and upper urinary tract; random cold-cup biopsies of the bladder and prostatic urethra, and complete transurethral resection of all bladder tumour visible on endoscopy, ensuring muscle is included in resected samples.
Drug: intravesical passive diffusion mitomycin — A dose of 40 mg mitomycin dissolved in 50 ml sterile water is infused intravesically through a Foley catheter, retained in the bladder for 60 min with catheter clamping, and then drained. Patients who have a complete response to the initial 6 weekly treatments underwent a further 10 monthly instillations, with the same dose and methods of infusion as initial assigned treatment.
  Other Names: Mitomycin-C
  Arms: Intravesical electromotive mitomycin; Intravesical passive diffusion mitomycin
Device: intravesical electromotive mitomycin — A dose of 40 mg mitomycin dissolved in 100 ml water is instilled and retained in the bladder for 30 minutes with 20 mA pulsed electric current, and then drained. Patients who have a complete response to the initial 6 weekly treatments underwent a further 10 monthly instillations with the same dose and methods of infusion as initial assigned treatment. Intravesical electromotive drug administration is given by a battery-powered generator delivering a controlled electric current that passes between the active intravesical electrode (integrated into a specific transurethral catheter) and dispersive ground electrodes (on skin of the lower abdomen). Operators set active electrode polarity and current intensity on the generator.
  Arms: Intravesical electromotive mitomycin

SUMMARY:
In laboratory and clinical studies, intravesical electromotive drug administration increased mitomycin bladder uptake, improving clinical efficacy in high-risk non-muscle invasive urothelial bladder cancer. The investigators' aim was to compare transurethral resection of bladder tumor and adjuvant intravesical electromotive mitomycin with transurethral resection and adjuvant intravesical passive diffusion mitomycin and transurethral resection alone in patients with primary stage pTa-pT1 and grade G1-G2 urothelial bladder cancer Patients will be randomly assigned to: transurethral resection alone, transurethral resection and adjuvant intravesical 40 mg passive diffusion mitomycin dissolved in 50 ml sterile water infused over 60 minutes once a week for 6 weeks, or transurethral resection and adjuvant intravesical 40 mg electromotive mitomycin dissolved in 100 ml sterile water with 23 mA pulsed electric current for 30 minutes once a week for 6 weeks. Patients in the intravesical adjuvant electromotive and passive diffusion mitomycin groups who are disease-free 3 months after induction treatment, will be scheduled to receive monthly intravesical instillation for 10 months, with the same dose and methods of infusion as initial assigned treatment. All patients will be assessed for safety. The investigators' primary endpoints are recurrence rate and disease-free interval. Analyses will be done by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven primary stage pTa-pT1 urothelial bladder cancer,
* adequate bone-marrow reserve (ie, white-blood-cell count ≥4000 × 10⁶ cells per L; platelet count ≥120 × 10⁹/L),
* normal renal function (ie, serum creatinine ≤123·76 μmol/L),
* normal liver function (ie, serum glutamic-oxaloacetic aminotransferase ≤42 U/L, serum glutamic-pyruvic aminotransferase ≤48 U/L, and total bilirubin ≤22 μmol/L),
* Eastern Cooperative Oncology Group performance status between 0 and 2.

Exclusion Criteria:

* non-urothelial carcinomas of the bladder;
* previous or concomitant grade G3 urothelial and/or carcinoma in situ of the bladder;
* urothelial carcinoma of the upper urinary tract and urethra, or both;
* previous intravesical treatment with chemotherapeutic and immunotherapeutic drugs;
* known allergy to mitomycin;
* bladder capacity less than 200 mL;
* untreated urinary-tract
* infection; severe systemic infection (ie, sepsis);
* treatment with immunosuppressive drugs;
* urethral strictures that would prevent endoscopic procedures and catheterisation;
* previous radiotherapy to the pelvis;
* other concurrent chemo therapy, radio therapy, and treatment with biological response modifiers;
* other malignant diseases within 5 years of trial registration (except for adequately treated basal-cell or squamous-cell skin cancer, in situ cervical cancer);
* pregnancy;
* any factors that would preclude study participation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 1994-01; Primary Completion 2004-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Disease-free interval | 120 months
  Time from randomisation to first cystoscopy noting recurrence as recorded by pathological assessment of transurethral-resection samples or biopsy samples

SECONDARY OUTCOMES:
Time to progression | 120 months
  time from randomisation until the onset of muscle invasive disease as recorded by pathological assessment of transurethral-resection samples or biopsy samples

OTHER OUTCOMES:
Overall survival | 120 months
  Time from randomisation until death from any cause
Disease-specific survival | 120 months
  Time from randomisation until death from bladder cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Savino M Di Stasi, MD, PhD, Principal Investigator — Tor Vergata University, Rome, Italy
Locations (1):
- Tor Vergata University, Department of experimental Medicine and Surgery/Urology, Rome, RM, Italy